CLINICAL TRIAL: NCT04908423
Title: Upper Extremity Injection of Xeomin® and Changes in Gait Related Mobility in Adults After Stroke
Brief Title: Xeomin® and Gait Related Mobility After Stroke
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00082738; BTX1.0 (Other: Atrium Health)
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: A one-group pretest-post-test experimental design will be used. Participants will be tested on the primary and secondary outcome measures before upper extremity injection with Xeomin® and 4 to 6 weeks thereafter.
Masking Description: To assess if Xeomin® injection into the hemiparetic arm is associated with changes in hemiparetic elbow range of motion, a blinded investigator will visually observe the position of the injected arm during their 10-meter walk test, using video tape sequences of the pre- and post-test gait analysis sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Xeomin® (Experimental): Participants will be injected via electromyographic guidance with a total of 200 units of Xeomin® into the pectoralis major, biceps brachii, brachioradialis, and latissimus dorsi muscles of the hemiparetic side using a standardized injection protocol (16). An additional 100 units of Xeomin® will be available at the discretion of the investigator for injection into additional affected upper extremity muscles
  Interventions: Drug: Xeomin®

INTERVENTIONS:
Drug: Xeomin® — To discover whether injection into the upper extremity with Xeomin® triggers improvements in gait-related mobility and quality of life in adults with hemiparesis secondary to stroke.
  Other Names: IncobotulinumtoxinA

SUMMARY:
The aim of the present pilot study is to evaluate the association between change in gait related mobility in ambulatory male and female adult hemiparetic patients before and 4-6-weeks after Xeomin® injection into the upper limb, using two standardized tests of physical function in outpatient rehabilitation that are widely used; the 10-meter walk test and the timed 'up and go' test (TUG).

DETAILED DESCRIPTION:
For this pilot study, the investigators hypothesize that there will be durational improvements in gait related mobility on the instrumented TUG and 10-meter walk tests 4-6-weeks post upper extremity Xeomin® injection. Physical function will be quantified as time to complete the instrumented TUG.

A one-group pretest-post-test experimental design will be used. Participants will be tested on the primary and secondary outcome measures before upper extremity injection with Xeomin® and 4 to 6 weeks thereafter. Additionally, participants will be contacted for an end of study visit via telephone approximately 12-weeks post Xeomin® injection to obtain information regarding any adverse events and gain insight into the therapeutic duration of the Xeomin®. The proposed duration of the study is 2 years to allow adequate time for screening, recruitment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiparesis and spasticity secondary to stroke with upper and lower limb spasticity and unilateral motor and/or sensory deficit
* No prior surgery to the lower limb
* Able to walk at least 10 meters without physical assistance from another person and without an assistive device
* Toe- ground clearance during swing phase without assistive device or orthoses
* No treatment with botulinum toxin within the past 4 months

Exclusion Criteria:

* Passive range of motion at either the ankle, knee, or elbow joint less than 30 degrees
* Participants with uncorrected hearing impairment
* Weight bearing restrictions due to concurrent orthopedic injuries that would make ambulating with or without an assistive device unsafe
* Speech language expression deficit (e.g., aphasia)
* Absence of proprioception upon neurologic examination
* Presence of fixed contractures in the upper or lower extremities not correctable to neutral
* Other confounding neurological diagnoses or active acute illness (cancer, Parkinson's disease, multiple sclerosis)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Instrumented Timed Up and Go test time | Baseline and 4-6 weeks after Xeomin injection
  Subjects arise from a chair, walk at their normal speed, turn around right after passing the tape at the end of the pathway, return to the chair, turn around and sit down. Subjects will be fitted with a , single Attitude and heading reference system (AHRS) sensor fixed on the manubrium inferior to the interclavicular notch in a chest-mounted pack. The AHRS is a wireless-telemetry, 10-parameter unit which includes a tri-axial accelerometer, a tri-axial gyroscope, a tri-axial magnetometer and an onboard temperature sensor.

SECONDARY OUTCOMES:
Change in Ten-meter walk test time | Baseline and 4-6 weeks after Xeomin injection
  Subjects walk 10-meters at self-selected pace
Change in Mini-Mental State Examination score | Baseline and 4-6 weeks after Xeomin injection
  Quantitative assessment of cognitive impairment. Scores range from 0-30, higher scores represent less cognitive impairment.
Change in Quality of Life in Neurological Disorders (Neuro-QoL) Depression - Short Form score | Baseline and 4-6 weeks after Xeomin injection
  Eight-item assessment of loss and feelings of hopelessness, negative mood, decrease in positive affect, information-processing deficits, negative views of the self, and negative social cognition in patients with neurological disorders. Scores range from 8-40, higher scores represent greater depressive symptoms.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) General Life Satisfaction - Short Form 5a score | Baseline and 4-6 weeks after Xeomin injection
  This form consists of 5-items and assesses the participant's cognitive evaluation of life experiences and whether that participant is content with their life. Scores range from 5-35, higher scores represent increased life satisfaction.
Change in Brief Pain Inventory (BPI) - Short Form score | Baseline and 4-6 weeks after Xeomin injection
  The BPI is a self-report measure that assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours. For the pain intensity portion of the assessment, scores range from 0-40, higher scores represent increased pain intensity. For the pain interference portion of the scale, scores range from 0-70, higher scores represent increased pain interference.
Change in Neuro-QoL Satisfaction with Social Roles and Activities - Short Form score | Baseline and 4-6 weeks after Xeomin injection
  A reliable and valid 8-item measure of involvement in social roles, activities and responsibilities. Scores for the social roles portion of the assessment range from 4-20, higher scores represent increased satisfaction with social roles. Scores for the activities portion of the assessment range from 4-20, higher scores represent increased activity satisfaction.
Change in Modified Ashworth Scale (MAS) score | Baseline and 4-6 weeks after Xeomin injection
  The MAS will be used as a measure of spasticity. Scores range from 0-4 for each muscle tested, higher scores represent increased spasticity.
Change in Berg Balance Scale (BBS) score | Baseline and 4-6 weeks after Xeomin injection
  The BBS is a 14-item objective tool that assesses static balance and fall risk in adults' post-stroke. Scores range from 0-56, higher scores indicate increased functional balance.
Change in Activities-Specific Balance (ABC) Scale score | Baseline and 4-6 weeks after Xeomin injection
  The ABC scale is a 16-item self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. Scores range from 0-100, higher scores indicate increased self-confidence with balance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Hirsch, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No